CLINICAL TRIAL: NCT01362803
Title: A Phase I/II Study of the Mitogen Activated Protein Kinase (MEK) 1 Inhibitor Selumetinib (AZD6244; Hydrogen Sulfate in Children With Neurofibromatosis Type 1 (NF1) and Inoperable Plexiform Neurofibromas (PN)
Brief Title: AZD6244 Hydrogen Sulfate for Children With Nervous System Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110161; 11-C-0161
Record Dates: First submitted 2011-05-27; First posted 2011-05-30 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-10-08

CONDITIONS: Neurofibromatosis 1; Neurofibromatosis Type 1; NF1; Neurofibroma, Plexiform
Keywords: Maximum Tolerated Dose; Pharmacokinetics; Pharmacodynamics; Response Rate; pain, quality of life and physical functioning
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Pain | interventions — AZD 6244

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Phase 1: AZD6244 PO BID x 28 DAYS
  Interventions: Drug: AZD6244
- Arm 2 (Experimental): Phase 2: AZD6244 PO BID x 28 DAYS
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — AZD6244 orally (at recommended Ph2 dose) every 12 hours on continuous daily schedule for cycles of 28 days until unacceptable toxicity, patient withdrawal or PD

SUMMARY:
Background:

- Plexiform neurofibromas are tumors that grow in and around nerves. The only way to treat them is with surgery. Some of these tumors cannot be completely removed. The tumors may be too large, too numerous, or in a bad location for surgery. An experimental drug called AZD6244 hydrogen sulfate may be able to prevent the tumors from growing, slow down their growth, or shrink them. This drug has been tested in adults with cancer and in children with some types of brain cancer. This study will test how well this drug works with these types of tumors.

Objectives:

- To study the safety and effectiveness of AZD6244 hydrogen sulfate in children and young adults with plexiform neurofibromas that cannot be completely removed by surgery.

Eligibility:

- Children and young adults between 12 and 18 years of age who have plexiform neurofibromas that cannot be completely removed by surgery.

Design:

* Patients will be screened with a physical exam, medical history, blood tests, and imaging studies.
* They will take the study drug twice a day with 8 ounces of water, every day for 28-day cycles of treatment. During study visits, participants will have blood and urine tests and physical exams. They will also have imaging studies to examine the tumor sizes and locations. They will answer questions about their health. They may have other tests as needed.
* Participants will continue to receive the study drug as long as they have no severe side effects and the disease is not getting worse.

DETAILED DESCRIPTION:
Background

* Patients with Neurofibromatosis 1 (NF1) have an increased risk of developing tumors of the central and peripheral nervous system, including plexiform neurofibromas (PN), which are benign nerve sheath tumors that are among the most debilitating complications of NF1. PN may be congenital and appear to have the fastest growth rate in young children. Surgery is the only standard treatment option available for PN. However, this is often difficult due to the encasement of vital structures, and extensive and invasive PN growth.
* PN are composed of neoplastic Schwann cells that lack NF1 gene expression. This results in upregulation of Ras, which initiates several signaling cascades regulating cell proliferation.
* Selumetinib (AZD6244 hyd sulfate), a novel orally bioavailable mitogen activated protein kinase inhibitor, is a specific inhibitor of MEK 1, which may mediate anti-tumor effects in PN by inhibition of downstream signaling of Ras. Selumetinib is currently undergoing evaluation in adult cancers and children with brain tumors.
* In this phase I study of selumetinib directed at NF1 PN, we have observed a degree of activity which has not been observed previously; therefore a phase II evaluation will be conducted.

Objectives

Phase I:

* To determine the maximum tolerated dose (MTD) of oral selumetinib administered daily to pediatric patients with NF1 and inoperable PN. Based on the results of the dose escalation in this study, the current MTD has been determined as 20 mg/m2/dose. To be consistent in pediatric dosing, an additional dose level of 25 mg/m2/dose was added, which is the MTD recently determined in a study conducted by the Pediatric Brain Tumor Consortium (PBTC). Amendment H (November 2014): The MTD has been determined to be 25 mg/m^2/dose.
* To define the acute and chronic toxicities and pharmacokinetics (PK) of selumetinib. Completed with amendment H.

Phase II:

-Primary objectives: To evaluate the confirmed partial and complete response rate of selumetinib using volumetric MRI analysis in children and young adults with NF1 and inoperable PN with PN related morbidity at the time of enrollment.

Eligibility

Pediatric Patients (>= 2 and <=18 years) who are able to swallow intact capsules, with NF1 and inoperable measurable PN that cause or have the potential to cause significant morbidity.

Design

* Selumetinib will be administered orally BID on a continuous dosing schedule (28 days = 1 treatment cycle). In the phase I portion, limited dose escalations will be performed to define the MTD based on tolerability of selumetinib during the first three treatment cycles. In the phase II portion, the recommended phase II dose level (RP2D) will be administered.
* Phase II: Patients will be enrolled on one of two strata:

  * Stratum 1: PN related morbidity present at enrollment

    ---PN related pain, disfigurement, or difficulty in physical functioning
  * Stratum 2: No significant PN related morbidity present at enrollment, but potential for development of PN morbidity
* Patient reported and functional outcomes will be evaluated at regular intervals.
* Disease status will be evaluated using volumetric MRI analysis at regular intervals.
* The day 1 and steady state plasma PK and PD of selumetinib will be evaluated.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age Phase I: >=3 years and <=18 years of age at the time of study enrollment, if able to swallow whole capsules. The age limits including young children were chosen because early childhood and puberty are considered to be the greatest risk for disease progression, and selumetinib may provide the most benefit to this young group of patients. In addition, an important objective of this study is to characterize the pharmacokinetics of selumetinib in the pediatric population since it has been well studied in adults.

   Age Phase II: >=2 and <= 18 years. BSA >= 0.55 m^2, and able to swallow whole capsules.
2. Diagnosis: Patients with NF1 and inoperable PN, defined as PN that cannot be surgically completely removed without risk for substantial morbidity due to encasement of, or close proximity to, vital structures, invasiveness, or high vascularity of the PN. The PN has to cause (stratum 1) or have the potential to cause (stratum 2) significant morbidity, such as (but not limited to) head and neck lesions that could compromise the airway or great vessels, paraspinal lesions that can cause myelopathy brachial or lumbar plexus lesions that could cause nerve compression and loss of function, lesions that could result in major deformity (e.g., orbital lesions) or are significantly disfiguring, lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions. Patients will be enrolled into stratum 1 or 2 based on PN related morbidity.

   Histologic confirmation of tumor is not necessary in the presence of consistent clinical and radiographic findings, but should be considered if malignant degeneration of a PN is clinically suspected.

   A PN is defined as a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches. A spinal PN involves two or more levels with connection between the levels or extending laterally along the nerve. In addition to PN, all study subjects must have either positive genetic testing for NF1 or have at least one other diagnostic criterion for NF1 listed below: (NIH Consensus conference):
   * Six or more cafe-au-lait macules (>=0.5cm in prepubertal subjects or >=1.5 cm in post pubertal subjects)
   * Freckling in axilla or groin
   * Optic glioma
   * Two or more Lisch nodules
   * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
   * A first-degree relative with NF1
3. Measurable disease: Patients must have at least one measurable PN, defined as a lesion of at least 3 cm measured in one dimension. Patients who underwent surgery for resection of a PN are eligible provided the PN was incompletely resected and is measurable.

   Phase II: Measurability and suitability for volumetric MRI analysis of the target PN must be confirmed with the NCI POB prior to enrolling a patient. The target PN will be defined as the clinically most relevant PN, which has to be amenable to volumetric MRI analysis. PN will be classified as "typical PN" versus "nodular PN" versus "solitary nodular PN" prior to enrollment
4. Prior Therapy: Patients with NF1 will only be eligible if complete tumor resection is not considered to be feasible without substantial risk or morbidity.

   * Since there is no standard effective chemotherapy for patients with NF1 and PN, patients may be treated on this trial without having received prior medical therapy directed at their PN.
   * Since selumetinib is not expected to cause substantial myelosuppression, there will be no limit to number of prior myelosuppressive regimen for PN or other tumor manifestations associated with NF1 such as optic glioma.
   * Patients who have received previous investigational agents or biologic therapy, such as tipifarnib, pirfenidone, Peg-Intron, sorafenib, imatinib or other targeted therapies are eligible for enrollment. At least 4 weeks must have elapsed since receiving medical therapy directed at the PN. Patients who received prior medical therapy for their PN must have recovered from the acute toxic effects of all prior therapy to <= grade 1 before entering this study.
   * Growth factors that support platelet or white cell number or function must not have been administered within the 7 days prior to enrollment.
   * At least 6 weeks must have elapsed prior to enrollment since the patient received any prior radiation therapy.
   * At least 4 weeks must have elapsed since any surgeries, with evidence of good wound healing.
5. Performance status: Patients >= 16 years of age must have a Karnofsky performance level of >=70%, and children <= 16 years old must have a Lansky performance of >=70%. Patients who are wheelchair bound because of paralysis secondary to a plexiform neurofibroma should be considered ambulatory when they are up in their wheelchair. Similarly, patients with limited mobility secondary to need for mechanical support (such as an airway PN requiring tracheostomy or CPAP) will also be considered ambulatory for the purpose of the study.
6. Hematologic Function: Patients must have an absolute neutrophil count >=1500/microliter, hemoglobin >=9g/dl, and platelets >=100,000/microliter.
7. Hepatic Function: Patients must have bilirubin within 1.5 x the upper limit of normal for age, with the exception of those with Gilbert syndrome, and AST/ALT within <= 3 x upper limit of normal.
8. Renal Function: Patients must have a creatinine clearance or radioisotope GFR >=60ml/min/1.73 m^2 or a normal serum creatinine based on age, described below.

   Age (years) / Maximum Serum Creatinine(mg/dL):

   Age <=5 / Maximum Serum Creatinine 0.8 mg/dL

   Age >5 to <=10 / Maximum Serum Creatinine 1.0 mg/dL

   Age >10 to <=15 / Maximum Serum Creatinine 1.2 mg/dL

   Age >15 / Maximum Serum Creatinine 1.5 mg/dL
9. Cardiac Function: Normal ejection fraction (ECHO or cardiac MRI) >= 53% (or the institutional normal; if a range is given then the upper value of the range will be used); QTC or QTcF <=450 msec.
10. Adequate Blood Pressure defined as:

    A blood pressure (BP) <= the 95th percentile for age, height, and sex measured. Adequate blood pressure can be achieved using medication for treatment of hypertension.
11. Informed Consent: Diagnostic or laboratory studies performed exclusively to determine eligibility for this trial must only be done after obtaining written informed consent from all patients or their legal guardians (if the patient is <18 years old). When appropriate, pediatric patients will be included in all discussions. This can be accomplished through one of the following mechanisms: a) the NCI POB screening protocol, b) an IRB-approved institutional screening protocol, or c) the study-specific protocol. Documentation of the informed consent for screening will be maintained in the patient s research chart. Studies or procedures that were performed for clinical indications (not exclusively to determine eligibility) may be used for baseline values even if the studies were done before informed consent was obtained.
12. Willingness to avoid excessive sun exposure and use adequate sunscreen protection if sun exposure is anticipated.
13. Willingness to avoid the ingestion of grapefruit and Seville oranges (as well as other products containing these fruits, e.g. grapefruit juice or marmalade) during the study, as these may affect selumetinib metabolism.

EXCLUSION CRITERIA:

1. Pregnant or breast-feeding females are excluded due to potential risks of fetal and teratogenic adverse events of an investigational agent. Pregnancy tests must be obtained prior to enrollment for all females of childbearing potential as per institutional standards (at NIH subjects 9 years and older or those showing pubertal development). Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Abstinence is an acceptable method of birth control.
2. Phase I: Patients who anticipate the need for surgical intervention within the first three cycles (3 months), as surgical intervention during the period of DLT evaluation may affect analysis of adherence and/or make the subject inevaluable.
3. Use of an investigational agent within the past 30 days.
4. Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumor, immunotherapy, or biologic therapy.
5. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses, or renal transplant, including any patient known to have hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) will be excluded. Patients with HIV who have adequate CD4 count, not requiring antiretroviral medication, may be enrolled.
6. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
7. Inability to swallow capsules, since capsules cannot be crushed or broken.
8. Inability to undergo MRI and/or contraindication for MRI examinations following the MRI protocol. Prosthesis or orthopedic or dental braces that would interfere with volumetric analysis of target PN on MRI.
9. Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
10. Prior treatment with selumetinib or another specific MEK1/2 inhibitor (unless the subject meets criteria for re-treatment).
11. Evidence of an optic glioma, malignant glioma, malignant peripheral nerve sheath tumor, or other cancer requiring treatment with chemotherapy or radiation therapy.
12. Supplementation with vitamin E greater than 100% of the daily recommended dose. Any multivitamin containing vitamin E must be stopped prior to initiation of therapy.
13. Patients not achieving adequate blood pressure in spite of antihypertensive therapy for control of blood pressure.
14. Cardiac Function:

    1. Known inherited coronary disease
    2. Symptomatic heart failure (NYHA Class II-IV prior or current cardiomyopathy, or severe valvular heart disease)
    3. Prior or current cardiomyopathy
    4. Severe valvular heart disease
    5. History of atrial fibrillation
15. Ophthalmologic conditions:

    1. Current or past history of central serous retinopathy
    2. Current or past history of retinal vein occlusion
    3. Known intraocular pressure (IOP) >= 21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of IOP). Patients with known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after discussion with the study chair.
    4. Subjects with any other significant abnormality on ophthalmic examination should be discussed with the Study Chair for potential eligibility
    5. Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbito-temporal PN (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
16. Known severe hypersensitivity to selumetinib or any excipient of selumetinib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib.
17. Recent major surgery within a minimum of 4 weeks prior to starting study treatment, with the exception of surgical placement for vascular access.
18. Any unresolved chronic toxicity with CTC AE grade >= 2 from previous anti-NF1 therapy, except for alopecia.
19. Clinical judgement by the investigator that the patient should not participate in the study.
20. While not an exclusion criterion, unless considered clinically indicated, patients should avoid taking other additional non-study medications that may interfere with the study medications. In particular, patients should avoid medications that are known to either induce or inhibit the activity of hepatic microsomal isoenzymes CYP1A2, CYP2C19 and CYP3A4, as this may interfere with the metabolism of selumetinib.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2011-09-21 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Ph2: Evaluate the confirmed partial and complete response rate of selumetinib in children and young adults with NF1 and inoperable PN. | prior to cycles 5,6,13,17,21,25 and then every 6 cycles
  Evaluate the confirmed partial and complete response rate of selumetinib in children and young adults with NF1 and inoperable PN.
Ph1: Determine MTD and extended tolerability | 3 treatment cycles
  Determine MTD and extended tolerability

SECONDARY OUTCOMES:
Study PK | first course
  pharmacokinetics (PK) of selumetinib at baseline and steady state
Ph2: Evaluate effect of selumetinib on bone mineral density, pain, quality of life and physical functioning. | before cycles 3,5,9,13 and then every 12 cycles
  DEXA, survey responses and functional evaluations
Ph2: Evaluate confirmed partial and complete response rate, and duration of response. | at each response evaluation
  Objective response rate
Ph2: determine long term tolerability, and safety | at each response evaluation
  Detailed clinical evaluation and laboratory studies
Measure adherence of chronic dosing | at each response evaluation
  level of adherence to selumetinib
determine effect on growth rate of PN | at time of PD
  Percent PN volume increase per year
Define toxicities | at each response evaluation
  describe and define the toxicities in pediatric patients on chronic dosing of selumetinib

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] Adeyemi A, Gross AM, Baldwin A, Dombi E, Widemann BC, Sint KJ. Selumetinib in pediatric patients with neurofibromatosis type 1 and plexiform neurofibroma: Propensity score analysis of SPRINT vs. natural history control arm. Neurooncol Adv. 2025 May 17;7(1):vdaf101. doi: 10.1093/noajnl/vdaf101. eCollection 2025 Jan-Dec. PMID 40709016
- [Derived] Gross AM, Achee C, Hart SE, Brewer L, Baldwin A, Wolters PL, Widemann BC; SPRINT study team. Selumetinib for children with neurofibromatosis type 1 and plexiform neurofibromas: A plain language summary of SPRINT. Future Oncol. 2024 May;20(14):877-890. doi: 10.2217/fon-2023-0565. Epub 2024 Feb 22. PMID 38869947
- [Derived] Gross AM, Dombi E, Wolters PL, Baldwin A, Dufek A, Herrera K, Martin S, Derdak J, Heisey KS, Whitcomb PM, Steinberg SM, Venzon DJ, Fisher MJ, Kim A, Bornhorst M, Weiss BD, Blakeley JO, Smith MA, Widemann BC. Long-term safety and efficacy of selumetinib in children with neurofibromatosis type 1 on a phase 1/2 trial for inoperable plexiform neurofibromas. Neuro Oncol. 2023 Oct 3;25(10):1883-1894. doi: 10.1093/neuonc/noad086. PMID 37115514
- [Derived] Gross AM, Glassberg B, Wolters PL, Dombi E, Baldwin A, Fisher MJ, Kim A, Bornhorst M, Weiss BD, Blakeley JO, Whitcomb P, Paul SM, Steinberg SM, Venzon DJ, Martin S, Carbonell A, Heisey K, Therrien J, Kapustina O, Dufek A, Derdak J, Smith MA, Widemann BC. Selumetinib in children with neurofibromatosis type 1 and asymptomatic inoperable plexiform neurofibroma at risk for developing tumor-related morbidity. Neuro Oncol. 2022 Nov 2;24(11):1978-1988. doi: 10.1093/neuonc/noac109. PMID 35467749
- [Derived] Gross AM, Wolters PL, Dombi E, Baldwin A, Whitcomb P, Fisher MJ, Weiss B, Kim A, Bornhorst M, Shah AC, Martin S, Roderick MC, Pichard DC, Carbonell A, Paul SM, Therrien J, Kapustina O, Heisey K, Clapp DW, Zhang C, Peer CJ, Figg WD, Smith M, Glod J, Blakeley JO, Steinberg SM, Venzon DJ, Doyle LA, Widemann BC. Selumetinib in Children with Inoperable Plexiform Neurofibromas. N Engl J Med. 2020 Apr 9;382(15):1430-1442. doi: 10.1056/NEJMoa1912735. Epub 2020 Mar 18. PMID 32187457
- [Derived] Dombi E, Baldwin A, Marcus LJ, Fisher MJ, Weiss B, Kim A, Whitcomb P, Martin S, Aschbacher-Smith LE, Rizvi TA, Wu J, Ershler R, Wolters P, Therrien J, Glod J, Belasco JB, Schorry E, Brofferio A, Starosta AJ, Gillespie A, Doyle AL, Ratner N, Widemann BC. Activity of Selumetinib in Neurofibromatosis Type 1-Related Plexiform Neurofibromas. N Engl J Med. 2016 Dec 29;375(26):2550-2560. doi: 10.1056/NEJMoa1605943. PMID 28029918
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0161.html